CLINICAL TRIAL: NCT04685213
Title: Electrical Stimulation Therapy for Preventing Hospital-acquired Weakness in Critically Ill COVID-19 Patients - A Proof of Concept Randomized Controlled Trial
Brief Title: Electrical Stimulation for Critically Ill Covid-19 Patients
Acronym: Phase I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Avazzia, Inc (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-47781-A
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Muscle Atrophy; Muscle Weakness
Keywords: electrical stimulation; skin perfusion; Muscle dysfunction
MeSH Terms: conditions — COVID-19; Muscular Atrophy; Muscle Weakness | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to intervention (IG) or control group (CG) with ratio of 1:1. The entire cohort will receive daily electrical stimulation (EE) in lower extremity (e.g. Gastronemius muscle) for up to 1 hour. The EE device will be functional for IG and non-functional for CG.
  Phase I will include patients (n=19) admitted to the hospital due to severe COVID-19 infection. The time frame for therapy will be 2 weeks or until hospital discharge, whichever comes first.
Who Masked: Participant, Care Provider
Masking Description: Devices may be active or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active E-Stim (Active Comparator): Subjects will receive an active electrical stimulation device to wear for 1 hour daily up to two weeks or until hospital discharge, whichever came first (phase I).
  Interventions: Device: Electrical Stimulation
- sham E-Stim (Sham Comparator): Subjects will receive a sham electrical stimulation device to wear for 1 hour daily up to two weeks or until hospital discharge, whichever came first (phase I).
  Interventions: Device: Electrical Stimulation - Sham

INTERVENTIONS:
Device: Electrical Stimulation — Subjects will receive an active electrical stimulation device to wear for 1 hour daily up to two weeks or until hospital discharge, whichever came first (phase I).
  Arms: Active E-Stim
Device: Electrical Stimulation - Sham — Subjects will receive a sham electrical stimulation device to wear for 1 hour daily up to two weeks or until hospital discharge, whichever came first (phase I).
  Arms: sham E-Stim

SUMMARY:
Unfortunately, hospital-acquired weakness is highly prevalent among COVID-19 hospitalized patients, who often require prolonged bed-rest or paralytics for an extended period of time in order to maintain oxygenation. Prolonged bed rest has been associated with pronounced loss of muscle mass that can exceed 10% over the 1st week, which leads to functional impairment and complications post-hospital discharge. Physical therapy and in-hospital mobility program may reduce the incident of hospital-acquired weakness, but they are often impractical for COVID-19 patients. In particular, conventional mobility programs are challenging for those who are being treated in an intensive Care Unit. The purpose of this study is to test feasibility and proof-of-concept effectiveness of daily use of lower extremity electrical stimulation (EE) therapy, as a practical solution to address lower extremity muscle deconditioning, to address chronic consequences of COVID-19 including hospital-acquired weakness.

DETAILED DESCRIPTION:
Phase I:

The purpose of this study is to test feasibility and proof-of-concept effectiveness of lower extremity electrical stimulation (EE) therapy to prevent muscular complications of COVID-19 including hospital-acquired weakness and neuropathy. This is a proof of concept randomized control trial (RCT) study for prevention. Eligible participants (n=19 anticipated) will be recruited from the Baylor St. Luke's' Medical Center (Houston, Texas). To be eligible participants should be hospitalized because of COVID-19 infection and suspected to be at risk for hospital acquired-weakness based on judgment of clinical intensivist investigators. Participants will be excluded if they are paralyzed. Other exclusion criteria include blow the knee amputation, those who have a demand-type cardiac pacemaker, implanted defibrillator or other implanted electronic device; those with wound infection, and other conditions that may interfere with outcomes or increase the risk of the use EE based on judgement of clinicians.

The Investigators hypothesize that implementation of EE as means of regular activation of lower extremity muscle is feasible and acceptable for the target population and would help to retain lower extremity muscle mass, lower extremity tissue oxygen saturation and perfusion, and thus reducing the severity of hospital acquired weakness and potentially improve outcomes of treatment among COVID-19 patients.

Participants will be randomized to intervention (IG) or control group (CG)). The entire cohort will receive daily EE in lower extremity (e.g. Gastronemius, tibial anterior muscle) up to 1 hour. EE therapy will be provided using a bio-electric stimulation technology (BEST) platform (Tennant Biomodulator PRO®, AVAZZIA, Inc.). The EE device will be functional for IG and non-functional for CG. The primary outcomes include between group difference and change from the baseline in muscle endurance, muscle strength, lower extremity tissue oxygen saturation, neuropathy, and muscle atrophy. Outcomes will be assessed at baseline, time of discharge or 2 weeks, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 test positive critically ill patients in need of assisted ventilation requiring care in the intensive care unit
* COVID-19 test positive critically ill patients in need of assisted ventilation requiring prolonged care in the hospital

Exclusion Criteria:

* Paralyzed patients (i.e., rocuronium, cisatracurium) at the moment of enrollment
* Patients under vasopressor therapy (i.e., norepinephrine, epinephrine, vasopressin) at the moment of enrollment
* Patients expected to be discharged in the next 24 hours
* Patient has a demand-type cardiac pacemaker, implanted defibrillator or other implanted electronic device.
* Active wound infection
* Below the knee amputations
* Based on the clinicians decision whether the patient is eligible for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Zulbaran-Rojas A, Mishra R, Rodriguez N, Bara RO, Lee M, Bagheri AB, Herlihy JP, Siddique M, Najafi B. Safety and efficacy of electrical stimulation for lower-extremity muscle weakness in intensive care unit 2019 Novel Coronavirus patients: A phase I double-blinded randomized controlled trial. Front Med (Lausanne). 2022 Dec 6;9:1017371. doi: 10.3389/fmed.2022.1017371. eCollection 2022. PMID 36561714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized into intervention (n=9), and control (n=10) groups.
Groups:
- Active E-Stim (Phase I): Subjects will receive an active electrical stimulation device to wear for 1 hour daily for up to 2 weeks.
- Sham E-Stim (Phase I): Subjects will receive a sham electrical stimulation device to wear for 1 hour daily for up to 2 weeks.
Period: Overall Study
Arm/Group | Active E-Stim (Phase I) | Sham E-Stim (Phase I)
Started | 9 | 10
Completed | 8 | 8
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active E-Stim (Phase I): Subjects enrolled in Phase I will receive an active electrical stimulation device to wear for 1 hour daily for up to 2 weeks.
- Sham E-Stim (Phase I): Subjects enrolled in Phase I will receive a sham electrical stimulation device to wear for 1 hour daily for up to 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Active E-Stim (Phase I) | Sham E-Stim (Phase I) | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (3.3) | 63.7 (2.9) | 65.8 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 2 | 1 | 3
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Gastrocnemius Muscle Endurance (Muscle Sustained Contraction) in Response to Electrical Stimulation
Description: Gastrocnemius muscle endurance in response to 5 minutes of electrical stimulation therapy will be assessed with surface electromyography using a validated non-invasive device (Delsys Trino Wireless EMG System, MA, US).
Time Frame: an average of 2 weeks (Phase I)
Measure: Mean (Standard Deviation); unit: milliVolts
Arm/Group | Active E-Stim (Phase I) | Sham E-Stim (Phase I)
Number analyzed (Participants) | 8 | 8
milliVolts | 352 (37) | 323 (18)

2. Primary Outcome: Change in Ankle Strength
Description: Ankle strength will be measured in response to the average of three 5-second dorsiflexion maximum voluntary isometric contractions per 30 seconds of relaxation in-between using a dynamometer (RoMech Digital Hanging Scale).
Time Frame: an average of 2 weeks (Phase I)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Active E-Stim (Phase I) | Sham E-Stim (Phase I)
Number analyzed (Participants) | 8 | 8
kg | 3.0 (1.6) | 2.1 (0.7)

3. Secondary Outcome: Change in Plantar Tissue Oxygen Saturation/Consumption
Description: Percentage of tissue oxygen saturation (SatO2) will be measured using a validated near-infrared (NIR) camera (Snapshot NIR, KENT Imaging Inc., Calgary, AB, Can) that detects an approximate value of real-time SatO2 level in superficial tissue. The metatarsus area including the five toes will be traced.
Time Frame: an average of 2 weeks (Phase I)
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Active E-Stim (Phase I) | Sham E-Stim (Phase I)
Number analyzed (Participants) | 8 | 8
Percentage of oxygen saturation | 69.2 (8.9) | 67.2 (9.5)

4. Other Pre Specified Outcome: Likelihood of Falling
Description: Assessment via the total score of Morse Fall Scale, which is the sum of six variables' score depending on presence or absence of:
  1. History of falling: Score 25 for falls during the present hospital admission or immediate history of physiological falls; if not, score 0.
  2. Secondary diagnosis: 15 if there is more than one medical diagnosis; if not, score 0.
  3. Ambulatory aids: 0 for walking without a walking aid, uses wheelchair, or is on bedrest; 15 for use of crutches, a cane, or a walker; 30 for ambulation clutching onto the furniture for support.
  4. Intravenous therapy: 20 for intravenous apparatus or a heparin lock inserted; if not, score 0.
  5. Gait: 0 if has a normal gait; 10 weak gait; 20 impaired gait.
  6. Mental status: patient's own self-assessment; 0 if normal; 15 if impaired.
  Scale:
  Minimum score or low risk: < 24 points Medium score or Moderate risk: 25-45 points Maximum score or high risk: > 45 points.
Time Frame: an average of 2 weeks (Phase I)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active E-Stim (Phase I) | Sham E-Stim (Phase I)
Number analyzed (Participants) | 8 | 8
score on a scale | 39.3 (11) | 46.2 (11.8)

5. Other Pre Specified Outcome: Change in Gastrocnemius Muscle Strength
Description: Gastrocnemius Muscle Strength will be assessed with surface electromyography using a validated non-invasive device (Delsys Trino Wireless EMG System, MA, US).
Time Frame: An average of 2 weeks (Phase I)
Measure: Mean (Standard Deviation); unit: milliVolts
Arm/Group | Active E-Stim | Sham E-Stim
Number analyzed (Participants) | 8 | 8
milliVolts | 6.5 (0.39) | 6.5 (0.36)

ADVERSE EVENTS:
Time Frame: an average of 2 weeks(phase I)
Description: Serious adverse events related to electrical stimulation therapy (e.g. pain, muscle damage, skin irritation) will be collected during the study.
Groups:
- Active E-Stim (Phase I): During Phase I of the study, four electrode pads will be placed in the proximal and distal gastrocnemius muscle of each participant in order to receive electrical stimulation therapy for 1 hour during hospitalization for an average of 2 weeks. Adverse events related to electrical stimulation therapy (i.e., pain, muscle damage, skin irritation) will be collected.
- Sham E-Stim (Phase I): During Phase I of the study, four electrode pads will be placed in the proximal and distal gastrocnemius muscle of each participant in order to receive electrical stimulation therapy for 1 hour during hospitalization for an average of 2 weeks. Adverse events related to electrical stimulation therapy (i.e., pain, muscle damage, skin irritation) will be collected. However, the sham group will receive an inactive device. So, electrical stimulation will only be provided to quantify the study outcomes. Adverse events will also be reported during this time.
Arm/Group | Active E-Stim (Phase I) | Sham E-Stim (Phase I)
All-Cause Mortality (participants affected / at risk) | 1/9 | 3/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT04685213/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT04685213/SAP_004.pdf
  • Informed Consent Form (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT04685213/ICF_002.pdf